CLINICAL TRIAL: NCT04932265
Title: Dissolution and Pharmacokinetic of Ginsenosides Released From Cyclodextrin Based Chewable Tablets: a Comparative, Randomized, Crossover, Open-label Study in Healthy Human Subjects.
Brief Title: Effect of Gamma-cyclodextrin on the Bioavailability of Ginsenosides
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Technical Problems with sensitivity of mass spectral detector
Sponsor: EuroPharma, Inc. (Industry)
Collaborators: Phytomed AB, Sweden (Unknown); Scientific Center of Drug and Medical Technologies Expertise of the Ministry of Health, Armenia (Unknown); CARDIOMED Family Health Center, LLC of the Ministry of Health of Armenia (Unknown); Institute of Fine Organic Chemistry of the National Academy of Science Yerevan, Armenia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EP-1008
Record Dates: First submitted 2021-06-01; First posted 2021-06-21 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Drug Absorption
Keywords: Ginsenosides Rg5; Ginsenosides Rk1; Compound K (CK).; Red ginseng HRG80; gamma-cyclodextrin; pharmacokinetic; relative bioavailability
MeSH Terms: interventions — gamma-cyclodextrin

STUDY DESIGN:
Intervention Model Description: A comparative study with the positive control, parallel groups, randomized, crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red ginseng HRG80 (Active Comparator): 16 subjects will receive 200 mg of red ginseng preparation HRG80 in one capsule
  Interventions: Dietary Supplement: HRG80™ Red Ginseng
- Red ginseng HRG80 incorporated in gamma-cyclodextrin (Experimental): 16 subjects will receive 200 mg of red ginseng preparation HRG80 incorporated in gamma-cyclodextrin in two chewable tablets
  Interventions: Combination Product: HRG80™ Red Ginseng + gamma cyclodextrin

INTERVENTIONS:
Dietary Supplement: HRG80™ Red Ginseng — Capsules containing red ginseng preparation HRG80 capsules, 200 mg - reference product
  Other Names: HRG80™ Red Ginseng Energy
  Arms: Red ginseng HRG80
Combination Product: HRG80™ Red Ginseng + gamma cyclodextrin — Chewable tablets containing red ginseng preparation HRG80 (100 mg) incorporated in gamma-cyclodextrin (GCD) - experimental modified product
  Other Names: HRG80™ Red Ginseng Energy Chewable
  Arms: Red ginseng HRG80 incorporated in gamma-cyclodextrin

SUMMARY:
This study will evaluate the relative bioavailability of ginsenosides Rg5, Rk1, and Ck of Red ginseng HRG80 preparations containing gamma-cyclodextrin (GCD) in the blood plasma of healthy subjects after oral administration of two different formulations of HRG80:

A. Capsules containing red ginseng preparation HRG80 (reference product) B. Chewable tablets containing red ginseng preparation HRG80 and GCD (modified product).

Dissolution testing measures the rate and extend water solubility of ginsenosides from the reference (A) and the modified (B) products. The difference of in vitro dissolution profiles between the reference (A) and modified (B) products will be assessed.

DETAILED DESCRIPTION:
A growing body of evidence suggests that gamma-cyclodextrin (GCD) can increase the clinical efficacy of water-insoluble biologically active compounds, which have low bioavailability. GCD is the most bio adaptable and applicable to increase the absorption of many drugs, including ginsenosides of Panax ginseng, by forming inclusion complexes or the form of GCD/drug conjugates. Ginsenosides have absolute bioavailability in the range from 0.2% to 48%, depending on the chemical structure and water solubility.

Hypothesis: gamma-cyclodextrin increases absorption and bioavailability of active constituents - Ginsenosides Rg5, Rk1, and Compound K (CK). The study aims to provide experimental evidence supporting or rejecting this hypothesis.

Sixteen healthy volunteers will be randomly assigned to receive two formulations, A and B, in two consecutive phases (Phase 1 and Phase) of an open-label study with a crossover design.

All patients will provide blood samples in each phase in each phase in 0.5, 0.75, 1, 2, 4, 6, 12, 24, and 48 hours (9 points) after drug administration, following will be a washout period for two weeks.

Subjects will be fasting for 10.00 hours before administering the investigational product. They will remain in the clinic post-dose until at least 24.00 hours each period, provided they are not suffering from any adverse event.

The concentration of ginsenosides Rg5, Rk1, and Ck in all blood samples will be determined using a validated analytical method (HPLC-MS) with the internal standard - digoxin. Appropriate mathematical methods and Kinetic 4.4.1 software will be used to generate basic pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, as determined by medical history, physical examination, and clinical laboratory testing,
* Willingness to stay in the unit overnight for the duration of the study,
* Provide a signed written informed consent.

Exclusion Criteria:

* overweight (BMI >35 kg/m2),
* pregnancy,
* lactation,
* drug abuse,
* use of dietary supplements or any form of medication (with the exception of oral contraceptives),
* heavy smokers, or ex-smokers with a remote history (> one pack/day),
* frequent alcohol consumption (>20 g ethanol/d),
* adherence to a restrictive dietary regimen,
* physical activity of more than 5 h/wk,
* respiratory tract infections, or suspicion thereof in the last 14 days before dosing,
* history or presence of disease in the kidneys and heart, lungs, liver, the gastrointestinal tract, endocrine organs, or other conditions such as the metabolic disease is known to interfere with the absorption, distribution, metabolism, and excretion of drugs,
* malignancy,
* autoimmune disorders such as (but not limited to) lupus erythematosus, multiple sclerosis, rheumatoid arthritis, or sarcoidosis,
* any other disease or condition, which, in the opinion of the Investigator, would make the subject unsuitable for this study,
* currently taking medications known to be CYP2C9 inducers (i.e., carbamazepine and rifampicin).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
The area under the plasma concentration versus time curve (AUC, expressed in ng x h/mL) of Rg5. | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The changes from the baseline the concentration (ng/ml) of Rg5 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
The area under the plasma concentration versus time curve (AUC, expressed in ng x h/mL) of Rk1. | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The changes from the baseline the concentration (ng/ml) of Rk1 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
The area under the plasma concentration versus time curve (AUC, expressed in ng x h/mL) of ginsenoside Ck | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The changes from the baseline the concentration (ng/ml) of ginsenoside Ck in blood plasma obtained after oral administration of the experimental product A or the active comparator B.

SECONDARY OUTCOMES:
The absorption rate constant (Ka, h-1) of Rg5 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The absorption rate constants (Ka, h-1) of Rg5 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
The absorption rate constant (Ka, h-1) of Rk1 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The absorption rate constants (Ka, h-1) of Rk1 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
The absorption rate constant (Ka, h-1) of Ck | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The absorption rate constants (Ka, h-1) of Ck in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Maximum plasma concentration (Cmax, ng/ml), of Rg5 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Maximum plasma concentration (Cmax, ng/ml), of Rg5 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Maximum plasma concentration (Cmax, ng/ml), of Rk1 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Maximum plasma concentration (Cmax, ng/ml), of Rk1 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Maximum plasma concentration (Cmax, ng/ml), of Ck | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Maximum plasma concentration (Cmax, ng/ml), of Ck in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Time to reach maximum plasma concentration, Tmax (h) of Rg5 . | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Time to reach maximum plasma concentration, Tmax (h) of Rg5 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Time to reach maximum plasma concentration, Tmax (h) of Rk1 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Time to reach maximum plasma concentration, Tmax (h) of Rk1 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Time to reach maximum plasma concentration, Tmax (h) of Ck. | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Time to reach maximum plasma concentration, Tmax (h) of Ck in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Mean absorption time MAT (h) of Rg5 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Mean absorption time MAT (h) of Rg5 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Mean absorption time MAT (h) of Rk1 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Mean absorption time MAT (h) of Rk1 in blood plasma obtained after oral administration of the experimental product A or the active comparator B.
Mean absorption time MAT (h) of Ck | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Mean absorption time MAT (h) of Ck in blood plasma obtained after oral administration of the experimental product A or the active comparator B.

OTHER OUTCOMES:
Relative bioavailability (%) of Rg5 incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Relative bioavailability (%) of Rg5 from 0 to 96 hours defined as the ratio of AUC0-96h for the tested formulation (B) to the AUC0-96h obtained for the reference product (A, 100%), given by the same route of administration in the same dose. F= AUCB/AUCA x 100%.
Relative bioavailability (%) of Rk1 incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Relative bioavailability (%) of Rk1 from 0 to 96 hours defined as the ratio of AUC0-96h for the tested formulation (B) to the AUC0-96h obtained for the reference product (A, 100%), given by the same route of administration in the same dose. F= AUCB/AUCA x 100%.
Relative bioavailability (%) of Ck incorporated in gamma-cyclodextrin | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  Relative bioavailability (%) of Ck from 0 to 96 hours defined as the ratio of AUC0-96h for the tested formulation (B) to the AUC0-96h obtained for the reference product (A, 100%), given by the same route of administration in the same dose. F= AUCB/AUCA x 100%.
Effect of gamma-cyclodextrin on absorption rate constant (Ka, h-1) of Rg5 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the absorption rate constants (Ka, h-1) of Rg5 obtained after oral administration of the experimental product A or the active comparator B.
Effect of gamma-cyclodextrin on absorption rate constant (Ka, h-1) of Rk1 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the absorption rate constants (Ka, h-1) of Rk1 obtained after oral administration of the experimental product A or the active comparator B.
Effect of gamma-cyclodextrin on absorption rate constant (Ka, h-1) of Ck | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the absorption rate constants (Ka, h-1) of Ck obtained after oral administration of the experimental product A or the active comparator B.
Effect of gamma-cyclodextrin on the maximal concentration (ng/ml) of Rg5 in blood | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the maximal concentration (ng/ml) of Rg5 obtained after oral administration of the experimental product A or the active comparator B.
Effect of gamma-cyclodextrin on the maximal concentration (ng/ml) of Rk1 in blood | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the maximal concentration (ng/ml) of Rk1 obtained after oral administration of the experimental product A or the active comparator B.
Effect of gamma-cyclodextrin on the maximal concentration (ng/ml) of Ck in blood | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the maximal concentration (ng/ml) of Ck obtained after oral administration of the experimental product A or the active comparator B.
the dissolution of Rg5 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the dissolution of Rg5 (% of the labeled content, Q) obtained in dissolution testing of the experimental product A or the active comparator B.
the dissolution of Rk1 | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the dissolution of Rk1 (% of the labeled content, Q) obtained in dissolution testing of the experimental product A or the active comparator B.
the dissolution of Ck | 0.5, 0.75, 1, 2, 4, 6, 12 and 24 hours, post-dose
  The difference in the dissolution of Ck (% of the labeled content, Q) obtained in dissolution testing of the experimental product A or the active comparator B.

CONTACTS AND LOCATIONS:
Overall Officials: Aghavni T Ginosyan, PhD, MD, Principal Investigator — Scientific Center of Drug and Medical Technologies Expertise of the Ministry of Health of the Republic of Armenia; Samvel Hairumyan, PhD, MD, Principal Investigator — CARDIOMED Family Health Center, LLC of the Ministry of Health of the Republic of Armenia; Areg Hovhannisyan PhD of A Hovhannisyan, Study Director — Institute of Fine Organic Chemistry of the National Academy of Science, Armenia
Locations (4):
- Armenia (3):
  - CARDIOMED Family Health Center, LLC of the Ministry of Health of the Republic of Armenia, Yerevan
  - Institute of Fine Organic Chemistry of the National Academy of Science, Yerevan
  - Scientific Center of Drug and Medical Technologies Expertise, Yerevan
- Phytomed AB, Våxtorp, HL, Sweden

REFERENCES:
- [Background] Yoo S, Park BI, Kim DH, Lee S, Lee SH, Shim WS, Seo YK, Kang K, Lee KT, Yim SV, Soung DY, Kim BH. Ginsenoside Absorption Rate and Extent Enhancement of Black Ginseng (CJ EnerG) over Red Ginseng in Healthy Adults. Pharmaceutics. 2021 Apr 2;13(4):487. doi: 10.3390/pharmaceutics13040487. PMID 33918329
- [Background] Zhou QL, Zhu DN, Yang YF, Xu W, Yang XW. Simultaneous quantification of twenty-one ginsenosides and their three aglycones in rat plasma by a developed UFLC-MS/MS assay: Application to a pharmacokinetic study of red ginseng. J Pharm Biomed Anal. 2017 Apr 15;137:1-12. doi: 10.1016/j.jpba.2017.01.009. Epub 2017 Jan 6. PMID 28086165
- [Background] Elshafay A, Tinh NX, Salman S, Shaheen YS, Othman EB, Elhady MT, Kansakar AR, Tran L, Van L, Hirayama K, Huy NT. Ginsenoside Rk1 bioactivity: a systematic review. PeerJ. 2017 Nov 17;5:e3993. doi: 10.7717/peerj.3993. eCollection 2017. PMID 29158964
- [Background] Kim HK. Pharmacokinetics of ginsenoside Rb1 and its metabolite compound K after oral administration of Korean Red Ginseng extract. J Ginseng Res. 2013 Oct;37(4):451-6. doi: 10.5142/jgr.2013.37.451. PMID 24235859
- [Background] Pan W, Xue B, Yang C, Miao L, Zhou L, Chen Q, Cai Q, Liu Y, Liu D, He H, Zhang Y, Yin T, Tang X. Biopharmaceutical characters and bioavailability improving strategies of ginsenosides. Fitoterapia. 2018 Sep;129:272-282. doi: 10.1016/j.fitote.2018.06.001. Epub 2018 Jun 5. PMID 29883635
- [Background] Quan LH, Jin Y, Wang C, Min JW, Kim YJ, Yang DC. Enzymatic transformation of the major ginsenoside Rb2 to minor compound Y and compound K by a ginsenoside-hydrolyzing beta-glycosidase from Microbacterium esteraromaticum. J Ind Microbiol Biotechnol. 2012 Oct;39(10):1557-62. doi: 10.1007/s10295-012-1158-1. Epub 2012 Jun 21. PMID 22717707
- [Background] Tannous M, Caldera F, Hoti G, Dianzani U, Cavalli R, Trotta F. Drug-Encapsulated Cyclodextrin Nanosponges. Methods Mol Biol. 2021;2207:247-283. doi: 10.1007/978-1-0716-0920-0_19. PMID 33113141
- [Background] Rivero-Barbarroja G, Benito JM, Ortiz Mellet C, Garcia Fernandez JM. Cyclodextrin-Based Functional Glyconanomaterials. Nanomaterials (Basel). 2020 Dec 15;10(12):2517. doi: 10.3390/nano10122517. PMID 33333914
- [Background] Li Z, Wang M, Wang F, Gu Z, Du G, Wu J, Chen J. gamma-Cyclodextrin: a review on enzymatic production and applications. Appl Microbiol Biotechnol. 2007 Nov;77(2):245-55. doi: 10.1007/s00253-007-1166-7. Epub 2007 Sep 22. PMID 17891389